CLINICAL TRIAL: NCT00772161
Title: A Single-Center, Single-Blind, Randomized, Oral Dose Cross-Over Study in Prepuberal Boys With ADHD to Investigate Efficacy and Bioequivalence of 20 mg Ritalin LA Compared to 20 mg Medikinet Retard After Treatment With o.d. Doses Over 7 Days Each.
Brief Title: Pharmacokinetics of Two Extended-Release Formulations of Methylphenidate in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: MPH-Kinetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Novartis (Industry)
Responsible Party: Prof. Dr. med. Eberhard Schulz, Universitätsklinik Freiburg
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRIT124DDE03; EudraCT Number: 2008-000227-25
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Disorder; Attention Deficit an Disruptive Behavior Disorders; Children; Central Nervous System Stimulants; Methylphenidate; Pharmacokinetics; Area Under Curve; Therapeutic Equivalency; Psychopharmacology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): First treatment week (day 1 to day 7) 20mg Ritalin LA; second treatment week (day 8 to day 14) 20mg Medikinet retard.
  Interventions: Drug: Methylphenidate
- Sequence 2 (Experimental): First treatment week (day 1 to day 7) 20mg Medikinet retard; second treatment week (day 8 to day 14) 20mg Ritalin LA.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Comparison of two extended-release formulations of 20mg Methylphenidate in a cross-over design.
  Other Names: Ritalin LA; Medikinet retard

SUMMARY:
This study is designed to provide pharmacokinetic data for the assessment of bioequivalence of Ritalin LA formulation compared to Medikinet ret. concerning plasma levels and efficacy measures.

The primary objective of the study is to determine the pharmacokinetic parameters and bioequivalence of Ritalin LA compared to Medikinet retard, both given as oral o.d. doses of 20 mg over 7 days in children with ADHD. The secondary objectives are to assess the efficacy, safety and tolerability of Ritalin LA and Medikinet retard and the association of these parameters with plasma levels.

DETAILED DESCRIPTION:
Study Design

This is a single center, Phase I, prospective, randomized, single blind, two-treatment cross-over study. 24 patients will be enrolled. Study duration for each patient is approximately 4 weeks (from screening/inclusion). Based on the assumption of 5 months recruitment, the total study duration will be approximately 6 month.

Target Population

A number of 24 prepubertal boys aged 8 - 14 years with Diagnosis of ADHD according to DSM IV will be enrolled in this study to ensure that 18 subjects will complete all assessments. The prepuberal status will be determined by Tanner stages ≤ 2. Diagnosis will be confirmed by the K-SADS-PL.

Patients will only be allowed to enter the trial if subject and subject´s parents/legal guardians provide informed consent about participation (following full explanation of the trial) and a written informed consent document is signed. In addition, it has to be verified by a physician that the patient meets all of the Inclusion Criteria and none of the Exclusion Criteria.

Study Treatment

Study medications will be either Ritalin LA 20 mg or Medikinet ret. 20 mg. Patients with a pre-treatment of psychotropic drugs other than Methylphenidate will have an individual washout period before inclusion to the study. This individual washout period will last 5 elimination half-life of the taken drug.

After randomization the patients will enter a 2 week treatment phase with a crossover at day 8. Patients randomized to Sequence 1 will be treated with Ritalin LA for the first week (day 1 to day 7) and with Medikiniet ret. for the second week (day 8 to day 14); patients randomized to Sequence 2 will be treated with Medikinet ret. for the first week (day 1 to day 7) and with Ritalin LA for the second week (day 8 to day 14). The study population will be randomized equally to the Sequence 1 or Sequence 2 group at Visit 2. The study ends 5 weeks after enrollment of the last patient (total study end).

ELIGIBILITY:
Inclusion Criteria:

* The patient and the parents/authorized legal representatives must understand the nature of the study and be able to comply with protocol requirements.
* Male patients aged 8-14 with Tanner stages 0 to 2 and a BMI between the 10th and 90th age percentile
* Patients having a diagnosis of ADHD of any type according to DSM-IV criteria, as established by history, psychiatric examination and a structured diagnostic interview (Kiddie-SADS-Present and Lifetime Version)
* Patients, whose symptoms are adequately controlled by a stable and well-tolerated dose of immediate release methylphenidate equivalent of 15 mg to 30 mg for at least one month before screening.
* Patients with parents or a legal guardian, who will give written informed consent for the child to participate in the study. Additionally, assent to participate must be obtained from all children entering the study. Assent will be documented by the child's signature on the consent form.
* Health status: Patients must have no clinically significant diseases or clinically significant abnormal laboratory values as assessed during medical history and physical exam.
* Patients meeting minimum intelligence requirements: In the opinion of the investigator the patient must generally be functioning at age-appropriate levels academically, which should take into account any prior cognitive or academic testing (basic knowledge of reading, writing and calculating).
* Patients already receiving behavioral therapies for ADHD may continue to do so during the course of the trial.

Exclusion Criteria:

* Patients with co-morbid psychiatric conditions with symptoms requiring current pharmacological treatment (e.g. major depression, psychosis).
* Patients with co-morbid psychiatric or somatic conditions that may contraindicate treatment or confound efficacy or safety assessments.
* Patients who are taking any concomitant medications likely to interfere with the study drug or confound efficacy or safety assessments, e.g. Tricyclic antidepressants, SSRIs except Fluoxetine, bupropion, clonidine, buspirone 2 weeks before randomization; Atomoxetine 2 weeks before randomization; Fluoxetine or antipsychotics 1 month before randomization; Pemoline and amphetamines 1 week before randomization.
* Patients with a known non-response to methylphenidate.
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.
* Patients who are judged by the investigator as likely to be non-compliant with study procedures, including those with a suspected history of substance abuse, or patients living with a person diagnosed with a substance abuse disorder.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Patients with warnings, mentioned in the German Basic Prescribing Information of Ritalin LA (SmPC in the current version) or Medikinet retard (SmPC in the current version): anorexia, severe depression, anxiety disorder, Gilles de la Tourette-Syndrome, other tic disorder, hypertension, occlusive arterial diseases, severe stenocardia, tachycardiac arrhythmia, stroke, hyperthyroidism, increased intra-ocular pressure, hypertrophy of the prostate, known hypersensitivity to sympathomimetics, MAO-inhibitors.
* Patients with a history of seizure disorder.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.

Ages: 8 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
C-max: Concentration of the Peak in the Plasma Concentration Curve | In Visit 3 (day 7) and Visit 4 (day 14): Repeated Assessment 1:00 h before and 0:30 h, 1:15 h, 2:15 h, 3:15 h, 4:15 h, 4:50 h, 5:30 h, 6:15 h, 8:00 h after medication intake
AUC-(0-inf): Area under the plasma concentration versus time curve extrapolated to infinity time | In Visit 3 (day 7) and Visit 4 (day 14): Repeated Assessment 1:00 h before and 0:30 h, 1:15 h, 2:15 h, 3:15 h, 4:15 h, 4:50 h, 5:30 h, 6:15 h, 8:00 h after medication intake

SECONDARY OUTCOMES:
Efficacy measure: SKAMP Combined rating, SKAMP-Attention subscale, SKAMP-Deportment subscale in a laboratory classroom setting. | In Visit 3 (day 7) and Visit 4 (day 14): Repeated Assessment at 0:25 h before and 0:50 h, 1:50 h, 2:50 h, 3:50 h, 5:50 h, 7:20 h after medication intake
Efficacy measure: Nisonger Child Behavior Rating Form - typical IQ Version (NCBRF-TIQ)from the primary caregiver. | Visite 2 ( Baseline, day 0), Visit 3 (day 7), Visit 4 (day 14)
Clinical Global Impressions - Severity of Illness scale (CGI-S) and Clinical Global Impressions - Improvement scale (CGI-I) by a child & adolescent psychiatrist | Visite 2 ( Baseline, day 0), Visit 3 (day 7), Visit 4 (day 14)
Assessment of Adverse Events | Visite 2 (Baseline, day 0), Visit 3 (day 7) and Visit 4 (day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fleischhaker, MD, Study Director — Universitätsklinikum Freiburg; Eberhard Schulz, Prof. Dr., Principal Investigator — Universitätsklinikum Freiburg; Klaus Hennighausen, MD, Study Chair — University Hospital Freiburg, Dep. for Child & Adoslecent Psychiatry
Locations (1):
- University Hospital Freiburg, Dep. for Child & Adolescent Psychiatry, Freiburg im Breisgau, Germany